CLINICAL TRIAL: NCT05750160
Title: The Effect of Music Therapy on Neutrophyl Lymphocytes Ratio, Interleukin 6 and Interleukin 10 Levels of Healthcare Workers With Burnout Syndrome
Brief Title: Music Therapy on Neutrophyl Lymphocytes Ratio, Interleukin 6 and Interleukin 10 Levels of Burnout Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yovita Mulyakusuma, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KET-1362/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2023-01-15; First posted 2023-03-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Burnout Syndrome; Neutrophil-Lymphocyte Ratio; Interleukin-6; Interleukin-10
MeSH Terms: conditions — Burnout, Psychological | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Given education only
- Intervention (Experimental): Given education and music therapy
  Interventions: Other: music therapy

INTERVENTIONS:
Other: music therapy — Music therapy that have been made by Music Therapist after Focus Group discussion, given three times a week for 4 weeks
  Arms: Intervention

SUMMARY:
Burnout Syndrome (BOS) can be defined as a state of stress both physically and psychically due to the burden and stressor of high work. The prevalence of BOS in health workers varies between 25-75% globally. Studies have shown that the presence of Burnout syndrome will meaningfully reduce the quality of services related to patient safety and cause immune system disorders that act as the body's defense against viral, bacterial, protozoal and fungal infections. Many strategies have been researched to help prevent and reduce the occurrence of Burnout syndrome, one of which is music therapy. The purpose of this study was to determine the effect of music therapy on the immune response in health workers with Burnout Syndrome.

This study is a randomized clinical trial with a pre and post test control group design for health workers at Dr Kariadi General Hospital and Dr. Cipto Mangunkusumo General Hospital. Subjects will be provided with information prior to the study and asked to sign an informed consent sheet if they agree to be involved in the study. Subjects will be divided into control groups and treatment groups with matching age, gender and type of work. In the treatment group, music therapy will be given as much as 3 times a week for 4 weeks. Data were taken on both groups before and after the intervention. This study used the Maslach Burnout Inventory Human Service Survey (MBI-HSS) and blood laboratory examination to determine the value of the Neutrophyl Lymphocyte Ratio, Interleukin 6 and Interleukin 10 levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years - 60 years old
2. Health workers in the wards and polyclinic of Dr. Cipto Mangunkusumo Hospital or Dr. Kariadi Hospital, including doctors in charge of patients, nurses, residents, and other supporting health workers
3. Included in the Burnout syndrome criteria from the Maslach Burnout Inventory-Human Service Survey questionnaire

Exclusion Criteria:

1. Refusing to follow the study
2. Have a history of heart disease, kidney disease, diabetes, cancer, tuberkulosis, autoimmune, immunodeficiency
3. Taking drugs that affect the central nervous system or immunosuppressants
4. Have hearing disorder
5. Have a psychiatric disorder
6. Being pregnant
7. Healthcare workers who don't like music

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Burnout syndrome | change from baseline score at 4 weeks
  Maslach Burnout Inventory Human Service Survey (MBI-HSS) score
Neutrophil Lymphocyte Ratio | Change from baseline Neutrophil Lymphocyte Ratio at 4 weeks
  Measured with Fluorescence Flow Cytometry
Interleukin 6 | Change from baseline Interleukin-6 level at 4 weeks
  Measured with Fluorescence Immunoassay
Interleukin 10 | Change from baseline Interleukin-10 level at 4 weeks
  Measured with ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Indonesia